CLINICAL TRIAL: NCT01173848
Title: A Randomized Study to Evaluate the Effectiveness of Cholecalciferol Versus Ergocalciferol Following Kidney Disease Outcomes Quality Initiative (K/DOQI) Guidelines for Vitamin D Therapy in Stages 3 & 4 Chronic Kidney Disease (CKD) Patients
Brief Title: Vitamin D Supplement Study for Stage Three and Four Chronic Kidney Disease (CKD) Patients
Acronym: UPGRADE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cleveland Clinic
Record Dates: First submitted 2010-07-30; First posted 2010-08-02 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2013-07

CONDITIONS: Chronic Kidney Disease Stage 3 and 4
Keywords: CKD; Vitamin D
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D2 (Active Comparator): Patients randomized to take vitamin D2
  Interventions: Drug: Ergocalciferol
- Vitamin D3 (Active Comparator): Patient's randomized to take Vitamin D3
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Ergocalciferol — 1.25mg weekly for 12 weeks then once a month for 3 months. or 1.25 weekly for 4 weeks then once a month for 5 months. or 1.25 monthly for 6 months
  Arms: Vitamin D2
Drug: Cholecalciferol — 1.25 weekly for 12 weeks then monthly for 3 months or 1.25 weekly for 4 weeks then monthly for 5 months or 1.25 monthly for 6 months
  Arms: Vitamin D3

SUMMARY:
The purpose of this study is to examine the effectiveness of vitamin D3 versus vitamin D2 in raising vitamin D levels and suppressing parathyroid hormone levels in patients with kidney disease who are not on dialysis.

DETAILED DESCRIPTION:
Subjects will be randomized and assigned to one of the treatment groups (D2 or D3). Subjects will be dispensed a supply of 1.25 mg cholecalciferol/ergocalciferol tablets, depending on their randomization outcome. The number of pills dispensed and medication instructions will be determined by their 25OHD level and K/DOQI guidelines. Both Study personnel and subject will be blinded to randomization group.

The treatment phase will be 24 weeks in duration with lab visits every 6 weeks. All laboratory specimens will be drawn either at CCF Main hospital labs or at a CCF family Health center lab. Subjects will be have telephone interviews at week 4, 10, 16, 22 and possibly at weeks 28 and 34.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years
* Chronic kidney disease stage 3-4 (eGFR 15-59 mL/min/1.73m2 body surface area, calculated using the MDRD Study equation GFR calculator)
* Hypovitaminosis D (serum 25OHD < 31 ng/mL)
* Secondary hyperparathyroidism (Intact PTH > 70 pg/mL for stage 3, and iPTH > 110 pg/mL for stage 4)

Exclusion Criteria:

* Initiation of vitamin D therapy between the time of the lab draw used for screening and the screening process
* History of liver failure
* History of intestinal malabsorption or chronic diarrhea
* Serum calcium level greater than 10.2 mg/dL
* Treatment with an activated vitamin D formulation (calcitriol, doxercalciferol or paricalcitol) within the past 6 months
* Treatment with phenobarbital, phenytoin, rifampicin, sucralfate, steroids, digoxin, or other medications that could affect vitamin D metabolism
* Primary hyperparathyroidism, active of a prior history of such
* Active malignancy excluding basal cell or localized squamous cell skin cancer
* Subject is pregnant (e.g. positive HCG test) or breast-feeding
* Refusal to use highly effective contraceptive measures (as determined by the investigator) throughout the treatment phase of the study
* Serum phosphorus level greater than 4.5 or treatment with an oral phosphate binder within the past 6 months
* Treatment with cinacalcet or other calcimimetic within the past 6 months
* Anticipated dialysis within 6 months after randomization
* Inability to swallow tablets
* Known sensitivity, intolerance, or other adverse response to the study drugs which would prevent compliance with study medication
* Have an unstable medical condition, defined as having been hospitalized within 30 days before screening, the expectation of recurrent hospital admissions or life expectancy of less than 6 months in the judgment of the investigator
* Subject is currently enrolled in, or fewer than 30 days have passed since subject has completed another investigational device or drug study(s); or subject is receiving another investigational agent(s).
* Current treatment with vitamin D 50,000 IU

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2011-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F Simon, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D2 | Vitamin D3
Started | 8 | 11
Completed | 4 | 3
Not Completed | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D2 | Vitamin D3 | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 5 | 8 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Subjects Achieving Normal Vitamin D Levels
Time Frame: within 24 weeks
Measure: Number; unit: participants
Arm/Group | Vitamin D2 | Vitamin D3
Number analyzed (Participants) | 8 | 9
participants | 4 | 4

ADVERSE EVENTS:
Groups:
- Vitamin D2 and Vitamin D3: Adverse Events were not logged by study arms.
  Patients randomized to take vitamin D2
  Ergocalciferol: 1.25mg weekly for 12 weeks then once a month for 3 months. or 1.25 weekly for 4 weeks then once a month for 5 months. or 1.25 monthly for 6 months
  or
  Patient's randomized to take Vitamin D3
  Cholecalciferol: 1.25 weekly for 12 weeks then monthly for 3 months or 1.25 weekly for 4 weeks then monthly for 5 months or 1.25 monthly for 6 months
Arm/Group | Vitamin D2 and Vitamin D3
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 7/19
Other Adverse Events (participants affected / at risk) | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D2 and Vitamin D3 (N=19)
Left Side Back Pain (Musculoskeletal and connective tissue disorders) | 1
Urinary Tract Infection (Endocrine disorders) | 1
Pneumonia (Infections and infestations) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Hospitalization (Infections and infestations) | 1
Acute Renal Failure (Endocrine disorders) | 1
Hospitalization for Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D2 and Vitamin D3 (N=19)
Nails Cracking and Falling Off (General disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Cystic Fibrosis (General disorders) | 1
Dizziness (General disorders) | 1
Worsening Hyperglycemia (General disorders) | 1
Cloudy Urine (Renal and urinary disorders) | 1
Hematuria (General disorders) | 1
Stomach Cramping (General disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
High Potassium (Metabolism and nutrition disorders) | 1
Urinary Tract Infection (Renal and urinary disorders) | 1
Allergies (General disorders) | 1
Leg Cramps (General disorders) | 1
Fatigue (General disorders) | 1
Acid Reflux (General disorders) | 1
Loose Stools (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
Adverse Events were not logged by study arms.

Early termination of the study lead to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes